CLINICAL TRIAL: NCT05126264
Title: Efficacy of the Dosage of a Non-steroidal Anti-inflammatory (Ibuprofen) on Inflammation and Postoperative Pain After Lower Third Molar Surgery.
Brief Title: Efficacy of Chronoterapy in Oral Surgery
Acronym: ECOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-000736-25
Record Dates: First submitted 2021-10-14; First posted 2021-11-18 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Tooth, Impacted; Trismus; Pain; Inflammatory Response
Keywords: Third molar; Chronotherapy; Ibuprofen; Randomized
MeSH Terms: conditions — Tooth, Impacted; Trismus; Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified dosage (Experimental): Ibuprofen pill at morning and afternoon; Placebo at night
  Interventions: Drug: Ibuprofen 400 mg
- Normal dosage (Active Comparator): Ibuprofen three times a day: morning, afternoon and night
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Ibuprofen 400 mg — morning and afternoon
  Other Names: Modified dosage
  Arms: Modified dosage
Drug: Ibuprofen 400 mg — morning, afternoon and night
  Other Names: Conventional dosage
  Arms: Normal dosage

SUMMARY:
Lower third molar extraction is one of the most common treatments in oral surgery practice. It is a treatment with inherent complications such as postoperative pain, swelling or trismus. In order to minimize disconfort after extraction, analgesic and anti-inflammatory medication is prescribed. Recently, it is seen that circadian rhythm may play an important role on drugs metabolism, modulating its effect depending on the moment of administration. The aim of the study is to analyze if dosage modification of a Non Steroideal Anti-Inflammatory (ibuprofen) affects on postoperative pain, swelling and open mouth limitation comparing to the normal dosage.

DETAILED DESCRIPTION:
A randomized crossover split-mouth clinical trial will be performed. After third molar extractions, patients will be prescribed ramdomly in one side wit the normal medication dosage while the contralateral side will be prescribed a modified dosage. Moreover, a blood sample will be obtained to analize the inflammatory profile.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years old
* Bilateral retained lower third molar

Exclusion Criteria:

* NSAID allergic
* Contraindication for surgical removal of third molar

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | From the day of the surgical procedure to the seventh-day
  Postoperative pain with visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain)

SECONDARY OUTCOMES:
Swelling | Baseline and post operatory (day 1, day 3, day 7)
  Distance from tragus to pogonion in milimiters

OTHER OUTCOMES:
Trismus | Baseline and post operatory (day 1, day 3 and day 7)
  Open mouth limitation in milimiters. Interincisal distance

CONTACTS AND LOCATIONS:
Locations (1):
- Fabian Perez Gonzalez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez-Corrales A, Campano-Cuevas E, Castillo-Dali G, Serrera-Figallo MA, Torres-Lagares D, Gutierrez-Perez JL. Relationship between salivary biomarkers and postoperative swelling after the extraction of impacted lower third molars. Int J Oral Maxillofac Surg. 2017 Feb;46(2):243-249. doi: 10.1016/j.ijom.2016.10.005. Epub 2016 Nov 3. PMID 27816275
- [Background] Albuquerque AFM, Fonteles CSR, do Val DR, Chaves HV, Bezerra MM, Pereira KMA, de Barros Silva PG, de Lima BB, Soares ECS, Ribeiro TR, Costa FWG. Effect of pre-emptive analgesia on clinical parameters and tissue levels of TNF-alpha and IL-1beta in third molar surgery: a triple-blind, randomized, placebo-controlled study. Int J Oral Maxillofac Surg. 2017 Dec;46(12):1615-1625. doi: 10.1016/j.ijom.2017.05.007. Epub 2017 Jun 10. PMID 28610818
- [Background] Keller M, Mazuch J, Abraham U, Eom GD, Herzog ED, Volk HD, Kramer A, Maier B. A circadian clock in macrophages controls inflammatory immune responses. Proc Natl Acad Sci U S A. 2009 Dec 15;106(50):21407-12. doi: 10.1073/pnas.0906361106. Epub 2009 Dec 1. PMID 19955445
- [Background] Curtis AM, Fagundes CT, Yang G, Palsson-McDermott EM, Wochal P, McGettrick AF, Foley NH, Early JO, Chen L, Zhang H, Xue C, Geiger SS, Hokamp K, Reilly MP, Coogan AN, Vigorito E, FitzGerald GA, O'Neill LA. Circadian control of innate immunity in macrophages by miR-155 targeting Bmal1. Proc Natl Acad Sci U S A. 2015 Jun 9;112(23):7231-6. doi: 10.1073/pnas.1501327112. Epub 2015 May 20. PMID 25995365